CLINICAL TRIAL: NCT04203524
Title: Impact of a Procalcitonin-Guided Algorithm on Antimicrobial Utilization in Critically Ill Cancer Patients with Sepsis: a Randomized Controlled Study (Pro-Can)
Brief Title: Procalcitonin and Antimicrobial Utilization in Critically Ill Cancer Patients with Sepsis
Acronym: Pro-Can
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No significant differences between 2 study arms
Sponsor: King Hussein Cancer Center (Other)
Responsible Party: Principal Investigator, Lama Nazer, Head of Pharmacy Research and Staff Development/ Critical Care Clinical Pharmacy Specialist, King Hussein Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 19KHCC11
Record Dates: First submitted 2019-12-14; First posted 2019-12-18 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-03

CONDITIONS: Sepsis; Septic Shock; Neoplasm; Critical Illness
Keywords: Procalcitonin; Sepsis; Septic shock; Cancer; Critical illness
MeSH Terms: conditions — Sepsis; Shock, Septic; Neoplasms; Critical Illness

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Procalcitonin Arm (Experimental): The medical team will be provided with a daily PCT for the patient, along with the PCT-guided algorithm that outlines the suggested management based on the PCT levels.
  Interventions: Diagnostic Test: Procalcitonin Levels
- Control Arm (Other): Procalcitonin levels will be measured for those patients, but the medical team will be blinded from their results
  Interventions: Other: Control

INTERVENTIONS:
Diagnostic Test: Procalcitonin Levels — Procalcitonin (PCT) will be measured within 48 hours of admission to the ICU or 48 hours of onset of sepsis (if developed during the ICU stay). In addition, the patients will have daily blood samples taken up to 5 days or until ICU transfer, whichever occurs first. A PCT-guided algorithm will be available to guide the management of patients in the PCT group.
  Arms: Procalcitonin Arm
Other: Control — Procalcitonin (PCT) will be measured within 48 hours of admission to the ICU or 48 hours of onset of sepsis (if developed during the ICU stay). In addition, the patients will have daily blood samples taken up to 5 days or until ICU transfer, whichever occurs first.The results of the PCT levels obtained will be blinded and all clinical team members will not be able to access the results.
  Arms: Control Arm

SUMMARY:
Studies have demonstrated that the use of a procalcitonin (PCT)-guided algorithm in combination with clinical judgment was associated with reduced antibiotic use without impacting mortality or treatment failure. Though several studies have evaluated the use of PCT in critically ill patients, there are limited studies that evaluated PCT in patients with cancer and many of the currently available studies have excluded immune-compromised patients.

This is a randomized controlled trial that aims to evaluate the impact of a procalcitonin-guided algorithm on antibiotic utilization in critically ill cancer patients with sepsis. In addition, the study aims to evaluate the predictive value of PCT for predicting mortality and positive cultures.

DETAILED DESCRIPTION:
Procalcitonin (PCT) has been widely studied to guide antibiotic use in critically ill septic patients. Using an algorithm for antibiotic de-escalation guided by PCT levels in septic patients with respiratory tract infections was associated with lower antibiotics exposure without increasing mortality or treatment failure. Furthermore, the current Surviving Sepsis Guidelines suggest that PCT levels may help clinicians in their decision of empiric antibiotics discontinuation especially in patients with suspected sepsis and low PCT values with no other evidence of infection (low level of evidence, GRADE 2C).

Reducing the use of antibiotics is a global health care priority. Using a PCT-guided algorithm in combination with clinical judgment was associated with reduced antibiotic use without increasing morbidity or mortality. Though PCT has been widely studied as a diagnostic, prognostic, and theragnostic inflammatory marker in patients with sepsis, there are limited studies that evaluated PCT in patients with cancer and many of the currently available studies have excluded immune-compromised patients. Furthermore, studies have reported elevated inflammatory markers, including PCT, in patients with cancer as a result of the malignancy itself or treatment complications. This may suggest that PCT alone may possibly be less useful for differentiating infectious from non-infectious sources of fever in cancer patients. However, serial PCT levels may be more useful in cancer patients, compared to a single level.

Sepsis is common in cancer patients; however, there are limited studies evaluating the clinical impact of obtaining PCT levels in this patient population. Therefore, this study will evaluate the impact of obtaining serial PCT levels on the number of antibiotic days in cancer patients with sepsis. In addition, the study aims to evaluate the predictive value of PCT for predicting mortality and positive cultures.

Study Objectives The main objective of this study is to evaluate the impact of a PCT-guided algorithm on the duration of antimicrobial therapy in critically ill cancer patients with sepsis. The main research question being asked is whether providing the clinical team with daily PCT levels, along with a PCT-based algorithm to guide antimicrobial management, would have an impact on the duration of antibiotic therapy. In addition, the study intends to assess the role of PCT in predicting mortality and positive cultures in the cancer septic patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Expected to remain in the ICU for at least 48 hours
* Patient meets the SEPSIS-3 criteria for sepsis defined as having a SOFA score change of 2 or more and suspected infection.
* Patient on antibiotics for suspected infection

Exclusion Criteria:

* Patient code is DNR
* Patient receiving antibiotics for surgical prophylaxis
* Consent cannot be obtained
* Patients who are expected to require antibiotics for more than 14 days
* Patients who have PCT levels ordered as part of their routine clinical care
* Patients who are followed by the Infectious Disease team.
* Patient with life expectancy <24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2019-08-21 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Time to antibiotic cessation | 28 days
  Time to antibiotic cessation at 28 days, hospital discharge, or death, whichever comes first after randomization
Number of antibiotic-free days | 28 days
  Number of antibiotic-free days at day 28 after randomization

SECONDARY OUTCOMES:
Antibiotic utilization | 28 days
  The antibiotic utilization will be evaluated by determining the antibiotic daily defined doses (DDD), as set by the World Health Organization, for each patient over the study period.

OTHER OUTCOMES:
Antibiotic de-escalation | 28 days
  Determined if de-escalation of antimicrobial therapy is performed during the ICU stay. De-escalation will be defined as reducing both the spectrum of antimicrobial therapy and its potential to promote resistance by driving selective pressure on microbiota. Reducing the number of antibiotics will also be considered as de-escalation.
Predictive value of PCT for both mortality | 28 days
  Determined by constructing a receiver operating characteristic (ROC) curve and the area under the ROC curve, as well as the sensitivity, specificity, and cut-off points with the highest predictability.
Recurrence of infection | 28 days
  Defined as a new infection that develops within 48 hours after stopping or de-escalating antibiotics.
Compliance with the PCT algorithm | 5 days
  The clinical decision of the medical team will be compared with the management suggested by the algorithm.
Predictive value of PCT for positive cultures | 28 days
  Determined by constructing a receiver operating characteristic (ROC) curve and the area under the ROC curve, as well as the sensitivity, specificity, and cut-off points with the highest predictability.

CONTACTS AND LOCATIONS:
Overall Officials: Lama H Nazer, PharmD, Principal Investigator — King Hussein Cancer Center
Locations (1):
- King Hussein Cancer Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shehabi Y, Sterba M, Garrett PM, Rachakonda KS, Stephens D, Harrigan P, Walker A, Bailey MJ, Johnson B, Millis D, Ding G, Peake S, Wong H, Thomas J, Smith K, Forbes L, Hardie M, Micallef S, Fraser JF; ProGUARD Study Investigators; ANZICS Clinical Trials Group. Procalcitonin algorithm in critically ill adults with undifferentiated infection or suspected sepsis. A randomized controlled trial. Am J Respir Crit Care Med. 2014 Nov 15;190(10):1102-10. doi: 10.1164/rccm.201408-1483OC. PMID 25295709
- [Background] de Jong E, van Oers JA, Beishuizen A, Vos P, Vermeijden WJ, Haas LE, Loef BG, Dormans T, van Melsen GC, Kluiters YC, Kemperman H, van den Elsen MJ, Schouten JA, Streefkerk JO, Krabbe HG, Kieft H, Kluge GH, van Dam VC, van Pelt J, Bormans L, Otten MB, Reidinga AC, Endeman H, Twisk JW, van de Garde EMW, de Smet AMGA, Kesecioglu J, Girbes AR, Nijsten MW, de Lange DW. Efficacy and safety of procalcitonin guidance in reducing the duration of antibiotic treatment in critically ill patients: a randomised, controlled, open-label trial. Lancet Infect Dis. 2016 Jul;16(7):819-827. doi: 10.1016/S1473-3099(16)00053-0. Epub 2016 Mar 2. PMID 26947523
- [Background] Schuetz P, Chiappa V, Briel M, Greenwald JL. Procalcitonin algorithms for antibiotic therapy decisions: a systematic review of randomized controlled trials and recommendations for clinical algorithms. Arch Intern Med. 2011 Aug 8;171(15):1322-31. doi: 10.1001/archinternmed.2011.318. PMID 21824946
- [Background] Andriolo BN, Andriolo RB, Salomao R, Atallah AN. Effectiveness and safety of procalcitonin evaluation for reducing mortality in adults with sepsis, severe sepsis or septic shock. Cochrane Database Syst Rev. 2017 Jan 18;1(1):CD010959. doi: 10.1002/14651858.CD010959.pub2. PMID 28099689
- [Background] Paul M, Dickstein Y, Raz-Pasteur A. Antibiotic de-escalation for bloodstream infections and pneumonia: systematic review and meta-analysis. Clin Microbiol Infect. 2016 Dec;22(12):960-967. doi: 10.1016/j.cmi.2016.05.023. Epub 2016 Jun 6. PMID 27283148
- [Background] Prkno A, Wacker C, Brunkhorst FM, Schlattmann P. Procalcitonin-guided therapy in intensive care unit patients with severe sepsis and septic shock--a systematic review and meta-analysis. Crit Care. 2013 Dec 11;17(6):R291. doi: 10.1186/cc13157. PMID 24330744
- [Background] Soni NJ, Samson DJ, Galaydick JL, Vats V, Huang ES, Aronson N, Pitrak DL. Procalcitonin-guided antibiotic therapy: a systematic review and meta-analysis. J Hosp Med. 2013 Sep;8(9):530-40. doi: 10.1002/jhm.2067. Epub 2013 Aug 17. PMID 23955852
- [Background] Wirz Y, Meier MA, Bouadma L, Luyt CE, Wolff M, Chastre J, Tubach F, Schroeder S, Nobre V, Annane D, Reinhart K, Damas P, Nijsten M, Shajiei A, deLange DW, Deliberato RO, Oliveira CF, Shehabi Y, van Oers JAH, Beishuizen A, Girbes ARJ, de Jong E, Mueller B, Schuetz P. Effect of procalcitonin-guided antibiotic treatment on clinical outcomes in intensive care unit patients with infection and sepsis patients: a patient-level meta-analysis of randomized trials. Crit Care. 2018 Aug 15;22(1):191. doi: 10.1186/s13054-018-2125-7. PMID 30111341